CLINICAL TRIAL: NCT02191332
Title: Collecting Data in Patients With HIV Infection Type 1 After Switching From a Protease Inhibitor-containing Therapy Regimen and a Viral Load Below Detection Level to a Viramune®-Containing Therapy Regimen
Brief Title: Observational Study in Patients With HIV Infection Type 1 After Switching to a Viramune®-Containing Therapy Regimen
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1305
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Viramune
  Interventions: Drug: Viramune

INTERVENTIONS:
Drug: Viramune

SUMMARY:
Observational study to collect data on maintaining anti-retroviral activity (quantitative HIV RNA determination) and immunological activity (CD4 cells) despite switching from protease inhibitor to nonnucleoside reverse transcriptase inhibitor (NNRTI) (Viramune®).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients with HIV type 1 infection

Exclusion Criteria:

* Counter-indications according to summary of product characteristics (SPC) for Viramune tablets
* No persons under 18
* Pregnancy and breast-feeding
* Use of oral contraceptives
* Use of drugs affecting CYP450 3A metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV treatment centres and HIV out-patient facilities
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 1999-12; Primary Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Change in viral load (HIV-RNA) | Baseline, after 26 and 52 weeks
Change in CD4 cell count | Baseline, after 26 and 52 weeks
Change in lipid status (lipodystrophy, triglycerides, cholesterol) | Baseline, after 26 and 52 weeks
  verbal rating scale
Change in glucose tolerance | Baseline, after 26 and 52 weeks
  verbal rating scale

SECONDARY OUTCOMES:
Assessment of subjective well-being | up to 52 weeks
  verbal rating scale
Assessment of tolerability by physician and patient | after 26 and 52 weeks
  verbal rating scale
Number of patients with adverse events | up to 52 weeks